CLINICAL TRIAL: NCT06134778
Title: Effect of Inspiratory Muscle Training on Cardiorespiratory Fitness, Pulmonary Function, Sports Skills, and Quality of Life in Wheelchair Rugby Athletes
Brief Title: Effect of Inspiratory Muscle Training on Cardiopulmonary Capacity in Wheelchair Rugby Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 40060714.5.0000.5235
Record Dates: First submitted 2023-10-26; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Breathing Exercises; Disability Physical; Athletes
Keywords: Inspiratory Capacity; Oxygen consumption; Spirometry; Exercise test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMT group (Experimental): Inspiratory muscle training group
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training was performed for six weeks. Athletes performed two daily sessions of 30 forced inspirations followed by long but not maximal expirations, with load adjusted between 50% and 60% of maximum inspiratory pressure, five times a week. A specific device was used for this purpose (Classic, Powerbreathe, United Kingdom), with light or medium resistance adjustment, depending on the subject's maximum inspiratory pressure.

SUMMARY:
The goal of this clinical trial is to learn about in inspiratory muscle training on cardiorespiratory capacity, pulmonary function, respiratory muscle strength, sports skills, and quality of life of wheelchair rugby athletes. The main question[s] it aims to answer are:

* Are the wheelchair rugby athletes show better results in cardiopulmonary assessment tests in safety and effort, in the post- inspiratory muscle training period, when compared to their results in the pre-inspiratory muscle training period?
* Is inspiratory muscle training capable of increasing ventilatory capacity at rest and during exertion?

Participants will be evaluated through questionnaires, laboratory and field tests, such as:

* Pulmonary function (spirometry),
* Inspiratory muscle strength (manovacuometry),
* Cardiorespiratory capacity under exertion (cardiopulmonary exercise test),
* Wheelchair rugby specific skills (Beck Battery)
* Quality of life (WHOQOL-DIS) .

DETAILED DESCRIPTION:
People with physical-motor disabilities, dependent on wheelchairs, have less mobility compared to people without disabilities, which can, in turn, have a direct and negative impact on the aerobic capacity and health of these individuals. Wheelchair Rugby (WCR) practitioners, as well as other sports, seek constant performance improvement, given the need to achieve better results in competitions. There has been an increase in the evaluation of parameters that may be related to better sports performance, as well as interventions that improve such performance. In relation to collective sports, such as WCR, the evaluation of important parameters such as maximum oxygen consumption during effort, maximum heart rate achieved and anaerobic limits, which enable adequate training adjustment, has gained prominence. Different interventions, such as inspiratory muscle training (IMT), aim to improve respiratory capacity and, consequently, cardiopulmonary capacity in savings and maximum effort. Therefore, this is a clinical study, with the objective of verifying the impact of IMT on cardiopulmonary performance, spirometric variables at rest and during effort, performance in field tests (Beck Battery) and quality of life in WCR athletes. Rugby athletes will be recruited in wheelchairs from teams in Rio de Janeiro, to perform two daily sessions of 30 forced inspirations followed by long, but not maximum, expirations, with a load adjusted between 50% and 60% of maximum inspiratory muscle strength, five times a week for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male gender,
* Age equal to or greater than 18 years,
* Presence of quadriplegia or tetra-equivalence,
* Wheelchair Rugby training time equal to or greater than six months,
* Participation in at least one official competition in the previous year the search.

Exclusion Criteria:

* The presence of musculoskeletal injury or pain that could interfere with the performance of movements in the wheelchair,
* Respiratory infections in the three weeks before the evaluations.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | Six weeks
  Using spirometry, in accordance with the recommendations proposed by the American Thoracic Society (Miller et al 2005). The variables considered were: absolute forced vital capacity and % of predicted, absolute forced expiratory volume in the first second and % of predicted, and absolute maximum forced expiratory flow and % of predicted, with measurement unit in liters (l).
Respiratory muscle strength | Six weeks
  Maximum inspiratory (MIP) and maximum expiratory pressures were evaluated using a digital manovacuometer (MVD300, MDI Produtos e Sistemas, Brazil) with measurement unit in CmH2O.
Cardiorespiratory capacity | Six weeks
  Cardiorespiratory fitness was assessed using the cardiopulmonary exercise test (CPET), performed on an upper limb cycle ergometer (Excite; TechnoGym; ITA). For the gas exchange analysis, a metabolic gas analyzer (Medical Graphics; VO2000; USA) was used. The variables peak oxygen consumption (VO2peak) (ml/kg/min), maximum effort time (min) and final load (w) were considered for analysis.

SECONDARY OUTCOMES:
Wheelchair Rugby specific skills | Six weeks
  The specific skills assessments of the WCR were performed through the application of the Beck Battery (Yilla & Sherril 1998; Gorla et al 2011) composed of the following tests: (i) passing accuracy; (ii) long-distance pass; (iii) ball-handling; (iv) blocking performance and (v) 20m speed.
Perceived quality of life | Six weeks
  For the quality of life assessment, participants completed the Brazilian version of the World Health Organization Quality of Life Questionnaire for People with Disabilities (WHOQOL-DIS) (Bredemeier et al 2014). The options for each item are described on a five-level Likert scale, where participants rate satisfaction from 1 to 5 (5 "totally agree" and 1 "totally disagree"). The results were presented on a scale of 0 to 100 (WHOQOL,1998), scaled in a positive direction. In other words, the higher the score, the greater the interviewee's perception of QoL in each domain (WHOQOL,1998).

OTHER OUTCOMES:
Sports training | Six weeks
  For the characterization of the study participants regarding injury and sports training, a questionnaire adapted from Gomes (2014) was applied, with questions related to WCR practice time, training routine, participation in competitions, functional classification, in addition to information about the type, level and time of injury.
Total body mass | Six weeks
  The measurement of total body mass (TBM) was carried out with the participant in his wheelchair, using a scale of adequate dimensions, with an accuracy of 0.1 kg (ID-M300/5, Filizola, Brazil) and measurement unit in kilogram (kg). To determine the final TBM, the weight of the wheelchair was discounted.
Height | Six weeks
  Height was measured with the participant in the supine position on a stretcher (tape measure with 0.1 cm precision; CESCORF, Rio Grande do Sul, Brazil) and measurement unit in centimeters (cm). The measurement of supine height was considered the distance between the plane of the vertex and the sole of the feet (Guedes & Guedes 2006).